CLINICAL TRIAL: NCT02716077
Title: Early FDG PET/CT Imaging as a Measure of Response in Patients With Melanoma on Pembrolizumab.
Brief Title: Early FDG PET in Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment due to changing treatment landscape for subject population
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: UPCC 11615
Record Dates: First submitted 2016-03-14; First posted 2016-03-23 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Clinical Stage III Nodal or Intransit Disease or Resectable Stage IV Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): FDG PET/CT scan pre-therapy
  Interventions: Radiation: FDG PET/CT imaging

INTERVENTIONS:
Radiation: FDG PET/CT imaging

SUMMARY:
Adult patients with histologically proven melanoma who will be treated with pembrolizumab will undergo FDG PET/CT scan as an early evaluation of response to therapy. Changes in FDG uptake will be correlated with lab and pathology results.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age
* History of histologically confirmed melanoma as assessed per medical record review.
* Eligible for the trial UPCC #01615, "A Phase Ib Tissue Collection Study of Pembrolizumab (MK-3475) in Subjects with Resectable Advanced Melanoma."
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine or serum pregnancy test at the time of the screening visit.
* Inability to tolerate imaging procedures in the opinion of the investigator or treating physician.
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.
* Ineligible for the trial UPCC #01615, "A Phase Ib Tissue Collection Study of Pembrolizumab (MK-3475) in Subjects with Resectable Advanced Melanoma."
* Only individuals (aged 18 or over) who can understand and give informed consent will be eligible to participate in this study. Individuals who are considered to be mentally disabled will not be recruited for this study. All subjects must be able to give informed consent. We will not be using specific methods to assess decisional capacity. Economically disadvantaged persons will not be vulnerable to undue influence, as this study offers no compensation. All individuals will be told that their choice regarding study participation will in no way change their access to clinical care. This should negate any undue influence or coercion. Children, fetuses, neonates, or prisoners are not included in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farwell, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States